CLINICAL TRIAL: NCT04830722
Title: A Randomized Single Center, Double Blinded, Split-body Clinical Trial of Poly-L-lactic Acid (Sculptra Aesthetic) for the Treatment of Cellulite of the Buttocks and Thighs
Brief Title: Clinical Trial of Poly-L-lactic Acid (Sculptra Aesthetic) for the Treatment of Cellulite of the Buttocks and Thighs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: Principal Investigator, Leslie Laser Aguilar, Regulatory Affairs Administrator, Goldman, Butterwick, Fitzpatrick and Groff
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sculptra-Aesthetic-2021
Record Dates: First submitted 2021-03-29; First posted 2021-04-05 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Cellulite
MeSH Terms: conditions — Cellulite

STUDY DESIGN:
Intervention Model Description: Enrolled subjects will be randomized to 2 treatment groups: "Right side treated" and "Left side treated". All subjects will receive three, single-sided injections of Sculptra Aesthetic, performed 1 month apart. Treatments will be provided to one side randomly assigned to either "right side" or "left side". The non-treatment side will receive bacteriostatic water, injected in the same manner as Sculptra Aesthetic.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Sculptra Aesthetic Side (Active Comparator): the treatment area side (an area side is considered either buttock and/or thigh) (left or right-depends on randomization) will receive up to two vials of Sculptra Aesthetic, for a total of 4 vials in one treatment session if 2 areas qualify.
  Interventions: Device: Sculptra Aesthetic
- Placebo side (Placebo Comparator): the treatment area side (an area side is considered either buttock and/or thigh) (left or right-depends on randomization) will receive 16 cc of bacteriostatic water, for up to 64 ccs of bacteriostatic water to match the volume injected on the active side
  Interventions: Device: Sculptra Aesthetic

INTERVENTIONS:
Device: Sculptra Aesthetic — One treatment side treated with Sculptra will be compared to the other side treated with bacteriostatic water (placebo) -same volume

SUMMARY:
clinical trial is to assess the safety, efficacy and patient satisfaction associated with the treatment of cellulite of the buttocks and thighs with injectable poly-L-lactic acid (PLLA), or Sculptra® Aesthetic

DETAILED DESCRIPTION:
Enrolled subjects will be randomized to 2 treatment groups: "Right side treated" and "Left side treated". All subjects will receive three, single-sided injections of Sculptra Aesthetic, performed 1 month apart. Treatments will be provided to one side randomly assigned to either "right side" or "left side". The non-treatment side will receive bacteriostatic water, injected in the same manner as Sculptra Aesthetic. Up to four (4) vials of Sculptra Aesthetic, diluted at 16 mL, will be used per treatment session.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult females age 30 to 60
* Both buttocks and/or both posterolateral thighs with a score of mild (1-5) to moderate (6-10 according to the Hexsel, Dal'Forno & Hexsel Cellulite Severity Scale (CSS), and a laxity score using the Hexsel, Dal'Forno & Hexsel Cellulite Severity Scale of 1 (slight) or 2 (moderate). Must be the same score on both sides of the same area (ie: if 1 on one buttock, must be 1 on the other buttock but can be a 2 on the thigh, as long as the other thigh is also a 2)
* Must be willing to give and sign an informed consent form and photographic release form.
* Must have had a stable body weight for at least 6 months prior to study entry.
* Must be willing to maintain usual sun exposure, diet, and exercise routines for the duration of the study.
* Subject agrees to avoid tanning or use of sunless tanner during the entire course of the study.
* Negative urine pregnancy test results at the time of study entry (if applicable).
* For female subjects of childbearing potential, must be willing to use an acceptable form of birth control during the entire course of the study. All systemic birth control measures must be in consistent use for at least 30 days prior to study enrollment participation.
* A female is considered of childbearing potential unless she is postmenopausal, without a uterus and/or both ovaries, or has had a bilateral tubal ligation.
* Acceptable methods of birth control are: oral contraceptives, contraceptive patches/rings/implants, Implanon®, Depo-Provera®, double-barrier methods (e.g. condoms and spermicide), abstinence and/or vasectomies of partner with a documented second acceptable method of birth control, should the subject become sexually activity.
* Must be willing to comply with study treatments and complete the entire course of the study.
* Cellulite that improves when the skin of the buttocks or thighs are stretched or distended superiorly.

Exclusion Criteria:

* Use of any of the following for the treatment of cellulite on either thigh or either buttock within the timelines identified below or intends to use any of the following at any time during the course of the study:
* Liposuction during the 12-month period prior to study treatment.
* Injections (eg, mesotherapy, dermal fillers, biostimulatory fillers, clostridium collagenase histolyticum); radiofrequency device treatments; laser treatment; buttock or thigh implant treatment; cryolipolysis; or surgery (including subcision and/or powered subcision) during the 24-month period before injection of study treatment.
* Any investigational treatment for cellulite on a buttock or thigh during the 12-month period before the injection of study treatment.
* Endermologie or similar treatments during the 6 month period before injection of study treatment.
* Massage therapy during the 3-month period before injection of study treatment.
* Creams (eg, Tretinoin, Celluvera™, TriLastin®) and/or home therapies to prevent or treat cellulite during the two week period before injection of study treatment.
* Subjects with scarring in treatment areas.
* Has any of the following local conditions in the areas to be treated (both buttocks or both thighs):
* History of lower extremity thrombosis or post-thrombosis syndrome.
* Vascular disorder (eg, varicose veins)
* A subject with tattoos or permanent implants in the treatment areas.
* A subject with history of or the presence of any skin condition/disease in the treatment area that might interfere with the diagnosis or evaluation of study parameters (i.e., atopic dermatitis, eczema, psoriasis).
* Subject who spray tanned or used sunless tanner in the treatment area 4 weeks prior to study treatment.
* A subject with an active bacterial, fungal, or viral infection in the treatment area.
* A subject with a significant history or current evidence of a medical, psychological, or other disorder that, in the investigator's opinion, would preclude enrollment into the study.
* Any history of bleeding or coagulation disorders.
* History of lidocaine sensitivity deemed by the investigator to preclude patient from enrolling in the study.
* A subject planning any other cosmetic procedure to the study treatment area during the study period, other than the treatment that will be performed by the investigator.
* Presence of incompletely healed wound in treatment area.
* Non-Ablative laser to the treatment area in the last 3 months.
* A female subject who is pregnant, nursing an infant or planning a pregnancy during the study.
* Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female adults age 30 to 60 who meet inclusion and exclusion criteria.
Enrollment: 20 (Estimated)
Dates: Start 2021-04-09 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Assessing Safety | 1 year
  Assessing safety of treatment of cellulite of the buttocks and thighs with injectable poly-L-lactic acid (PLLA), or Sculptra® Aesthetic (Galderma Laboratories, Fort Worth, TX) using Evaluation of side effects by subject and investigator
Assessing Efficacy | 1 year
  Assessing efficacy of treatment of cellulite of the buttocks and thighs with injectable poly-L-lactic acid (PLLA), or Sculptra® Aesthetic (Galderma Laboratories, Fort Worth, TX) using Subject and Blinded Investigator GAIS and Blinded Investigator Hexsel Grading Scale, Galderma Cellulite Grading Scale, and end of study iodentification of correct treatment side using side by side photography before unblinding.
Assessing Patient Satisfaction | 1 year
  Assessing patient satisfaction of treatment of cellulite of the buttocks and thighs with injectable poly-L-lactic acid (PLLA), or Sculptra® Aesthetic (Galderma Laboratories, Fort Worth, TX) using a patient satisfaction questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Fabi, MD, Principal Investigator — Cosmetic Laser Dermatology
Locations (1):
- Cosmetic Laser Dermatology/West Dermatology Research Center, San Diego, California, United States

REFERENCES:
- [Background] Haddad A, Menezes A, Guarnieri C, Coimbra D, Ribeiro E, Sarubi J, Avelar LE, Del Nero MP, da Cunha MG, Mazzuco R, Kamamoto C, Cazerta C. Recommendations on the Use of Injectable Poly-L-Lactic Acid for Skin Laxity in Off-Face Areas. J Drugs Dermatol. 2019 Sep 1;18(9):929-935. PMID 31524350
- [Background] Narins RS, Baumann L, Brandt FS, Fagien S, Glazer S, Lowe NJ, Monheit GD, Rendon MI, Rohrich RJ, Werschler WP. A randomized study of the efficacy and safety of injectable poly-L-lactic acid versus human-based collagen implant in the treatment of nasolabial fold wrinkles. J Am Acad Dermatol. 2010 Mar;62(3):448-62. doi: 10.1016/j.jaad.2009.07.040. PMID 20159311
- [Background] Jabbar A, Arruda S, Sadick N. Off Face Usage of Poly-L-Lactic Acid for Body Rejuvenation. J Drugs Dermatol. 2017 May 1;16(5):489-494. PMID 28628686
- [Background] Davis DS, Boen M, Fabi SG. Cellulite: Patient Selection and Combination Treatments for Optimal Results-A Review and Our Experience. Dermatol Surg. 2019 Sep;45(9):1171-1184. doi: 10.1097/DSS.0000000000001776. PMID 30913048
- [Background] Uebel CO, Piccinini PS, Martinelli A, Aguiar DF, Ramos RFM. Cellulite: A Surgical Treatment Approach. Aesthet Surg J. 2018 Sep 14;38(10):1099-1114. doi: 10.1093/asj/sjy028. PMID 29432568
- [Background] Mazzuco R, Sadick NS. The Use of Poly-L-Lactic Acid in the Gluteal Area. Dermatol Surg. 2016 Mar;42(3):441-3. doi: 10.1097/DSS.0000000000000632. No abstract available. PMID 26859651
- [Background] Lin MJ, Dubin DP, Khorasani H. Poly-L-Lactic Acid for Minimally Invasive Gluteal Augmentation. Dermatol Surg. 2020 Mar;46(3):386-394. doi: 10.1097/DSS.0000000000001967. PMID 31188150
- See also: Accessed September 18th 2020 — http://www.accessdata.fda.gov/cdrh_docs/pdf3/P030050S002c.pdf